## **Cover Page:**

ClinicalTrials.gov#: NCT03880032

**IRB Approved Consent Document:** Biological Supplement Study Consent

Title: Happy Mother-Healthy Baby: An Anxiety-focused Early Prenatal Intervention -

Biological Supplement Study

**Document Date:** July 25, 2019

## HAPPY MOTHER. HEALTHY BABY STUDY-BIOLOGICAL SUBSTUDY

Main Consent to Participate in the SubStudy

## (This consent statement must be read (prior to Baseline Data Collection) to those women who screen eligible and are interested in participating in the study)

<u>Introduction:</u> As-salaam-u-alaikum. Thank you for your interest in our new program, "Happy Mother, Healthy Baby" (HMHB). We are conducting research to learn if HMHB can improve maternal well-being and child health at Holy Family Hospital. Before you decide to take part in this research, you need to know the purpose of this program and what it will involve.

The purpose of the Happy Mother Healthy Baby Research Project: Many mothers feel stressed, nervous, or anxious during pregnancy. The purpose of this research is to learn if our HMHB program can reduce this anxiety and improved their wellbeing. This could help the health of both the mother and her baby. If you participate, we will ask your permission to also collect information about your baby's health. In addition, we are trying to understand the causes of anxiety in pregnant and postpartum women; to do so we will be collecting blood.

Why are we requesting your participation in this program?: We want to include about 1200 pregnant mothers like you from Rawalpindi who are over 18 years old. It is important that we gather information from women who show some signs of being anxious and some women who don't in order to compare them. Mothers who agree to participate and do not show signs of anxiety will be put in the routine care group. Mothers who agree to participate and show signs of anxiety will be divided into two groups, the Routine Care group and the HMHB group. If you are put in the Routine Care group, hospital staff will help you with issues related to your health or your baby's health, when you come for up to 8 antenatal care visits. They are trained to help you with any mental health concerns you might have, such as feeling anxious. You will also be reimbursed for your transportation to come to these antenatal visits and for the costs ultrasounds indicated by your providers at Holy Family Hospital.

• If you are in the HMHB group, you will receive this same help from hospital staff, and also participate in the HMHB intervention. Our intervention includes six main sessions plus up to six additional sessions, if needed, that will focus on managing stress while you are pregnant. The number of the six additional sessions will depend on your stage of pregnancy when you enroll. Each session will be done here with our project staff, will last about 45 minutes, and will focus on specific goals for improving your health and your child's health. Your family will be invited to participate in three sessions to facilitate your getting their support. As in the Routine Care group, you will also be reimbursed for your transportation to come to these antenatal visits and for the costs of ultrasounds indicated by your providers at Holy Family Hospital.

<u>Can I choose which group I want to be in?</u>: No. We will use a computer program to put you in one of the groups, with an equal chance of being in either of the two groups, like tossing a coin. The researchers, who ask you questions and analyze the information, will not know which group you are in. Only the hospital staff and research team members at the hospital will know. This will help make sure that the findings are not affected by this information.

What data will we collect? Participation in the study depends on your allowing us access to your chart to record information about the pregnancy, the growth of your baby, and about medical conditions and medications. In addition to data we collect during your participation in routine antenatal care visits (group 1) or the HMHB sessions (group 2), we will also collect some information at four different times. I will describe these now, referring to them as "Start of Study Visit", "Late Pregnancy Visit", "Delivery/Birth Visit", and "End of Study Visit". Questions at some of the visits will

HMHBSupp - Form S001 - Main Study + Substudy Consent - July 25, 2019

refer to sensitive topics. We will also analyse blood that is collected by your doctors or a trained member of our study staff to examine changes in your hormones, inflammation, and other biological functions during pregnancy. This will be done at the first study visit, in the 2<sup>nd</sup> trimester, and in the 3<sup>rd</sup> trimester. We will also collect a final blood sample at the end of study visit at 6 weeks postpartum. Specifically, in terms of other information we will be asking you about or gathering from your records:

- At the Start of Study Visit we will ask you about some demographic information (like your age, years of education), about your mood, stress you are feeling, your relationships with others, any health problems you have experienced recently, medication you may be taking, and/or any care you might have sought. We will also draw your blood. This visit will take about 1 hour.
- At a second trimester visit, we will ask you questions about your mood and anxiety and will draw your blood.
- At the Late Pregnancy Visit we will ask you about your mood and anxiety as well as any stress or nervousness you may be feeling in general or related to the pregnancy, the support you receive, the nature of your relationships, daily functioning, and use of medical services during your pregnancy. We will also access your chart and record information about pregnancy conditions, the growth of your baby (from ultrasound), and about medical conditions and medications. We will also draw your blood. The interview done to collect this information will take about 1 hour and will be done during one of your already scheduled visits.
- The *Delivery/Birth Visit* will be done as soon as possible after your delivery. We will only ask
  you a few questions about breastfeeding; these will take about 5 minutes. We will also access
  at your chart and record information about your labor and delivery, the care your received, and
  some information about your baby, like the weight and size.
- The *End of Study Visit* will be completed at your 6-week postpartum visit here at the hospital. At that time, we will do another interview, again asking you questions about stress, whether you feel anxious or down, the support you receive, the nature of your relationships, daily functioning, adverse events you may have experienced, breastfeeding of your infant, and use of medical services during your pregnancy. Other questions will include things like how confident you feel in taking care of your baby and of taking actions, and how close you feel to your baby. As with the other visits, we will also access your chart to record information about the pregnancy, the growth of your baby, and about medical conditions and medications. We will also draw your blood. Finally, we will administer a scale to assess the development of your baby. This visit will take up to two hours. If the results of the scale indicate that your baby is at risk of later developmental delays, we will re-contact you after completion of the study to give you this information and explain the test results with you.
- Throughout the study we will access yours and your child's medical records when needed to get information about the health of you and your baby.

<u>Do I have to take part?</u>: No, you do not have to take part in this program, participation is voluntary. You have a right to withdraw at any time without giving any reason, without penalty or loss of benefits to which you are otherwise entitled. Refusing to take part will not result in any penalty or loss of benefits.

What are the possible benefits of taking part?: By participating in this program, mothers may be able to lower their level of anxiety. The program will also help mothers notice feeling nervous and deal with it so that it is less likely to harm her or her infant. The information you will provide taking part in the study will help us to improve maternal and child health services. This study may also help

HMHBSupp - Form S001 - Main Study + Substudy Consent - July 25, 2019

us to understand biological mechanisms underlying anxiety during pregnancy. Another benefit will be reimbursement for medically indicated ultrasounds during your prenatal care.

What are the possible disadvantages and risks of taking part?: We will be asking you questions at several points in time. This may take an hour of your time at each session and answering may make you tired. Also, talking about your feelings can sometimes be difficult and might make you upset. If you feel stressed, you will be offered to speak to a counselor. You can refuse to answer any questions that you are not comfortable answering. You also have the right to stop the interview at any time if you feel unhappy. A blood draw can include temporary discomfort, bleeding or bruising, and rarely infection and light-headedness/fainting. Whenever possible, we will plan to use blood collected from the blood draws that your health care provider is already requesting during pregnancy, so that you will not need an additional blood stick.

<u>Payment for participation:</u> You will not receive any payment. However, you will be reimbursed for transportation costs for the study visits and the costs of ultrasounds needed for your prenatal care, if you choose to take part. You will also receive a gift at the conclusion of the study in the form of gifts for the baby.

<u>Will my information be kept confidential?</u>: All information that we collect from you will be kept confidential and safe. This includes the information you tell us and any information about you or your baby that we copy from your medical records. Although the information from the surveys is confidential, if you are at risk of hurting yourself or your child—including infant neglect or abuse -- it is the legal and ethical responsibility of the research team to share that information with others. We will ask your permission before your information is shared with your health care providers.

<u>Who approved this study?</u>: The Ethical Review Board of Rawalpindi Medical University and the Ethical Review Board of Johns Hopkins University have approved this study. This research is funded by the National Institutes of Mental Health in the United States. This study is protected by a Certificate of Confidentiality that helps keep your information private when stored in the US.

Who I can contact in case of complaints?: To learn more about this study, you can call the phone numbers provided at the end of this information sheet at any time Monday to Friday, from 9AM to 5 PM.

Gynaecology and Obstetrician Department

Phone number: xxxxxxx

## What do I do to participate?

If you agree to take part in this study, you will be asked to sign or put a thumb impression on the consent form. You must answer 'yes' and initial to all four questions in the boxes below in order to enroll in the study.

| Name of person taking consent: | | |
|---|---|---|
| | Plea | se initial all boxes |
| 1. | I confirm that I have understood the information in the attached document. I have had the chance to carefully consider it and ask questions. I was provided with satisfactory replies for my questions. | |

| нмнвя | Supp - Form S001 – Main Study + Substudy | Consent — July 25, 2019 | |
|---|---|---|---|
| 2. | I understand that my participation is entirely voluntary. I am free | | |
| | to withdraw at any time with | / decision to | |
| | withdraw from the study will i | that I receive | |
| | or my legal rights. | | |
| 3. | I understand that the informati | idential. I also | |
| | give permission to the research | | |
| | with HMHB study to access i | | |
| 4. | from medical records, when not agree to take part in the stud | | |
| т. | ragice to take part in the stud | | |
| Name of participant | | Date | Signature |
| , , | | | J |
| | | | ••••• |
| ii the | participant is unable to provide | a signature above. | |
| Name of witness | | Date | Signature |
| | | 24.0 | 3191141413 |
| Name of person taking consent | | Date | Signature |